CLINICAL TRIAL: NCT00002703
Title: A PHASE III TRIAL EMPLOYING CONFORMAL PHOTONS WITH PROTON BOOST IN EARLY STAGE PROSTATE CANCER: CONVENTIONAL DOSE COMPARED TO HIGH DOSE IRRADIATION
Brief Title: Radiation Therapy in Treating Patients With Stage I or Stage II Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Proton Radiation Oncology Group (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000064503; PROG-9509
Record Dates: First submitted 1999-11-01; First posted 2004-09-01 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2012-04

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

INTERVENTIONS:
Radiation: high-LET heavy ion therapy
Radiation: low-LET photon therapy

SUMMARY:
RATIONALE: Radiation therapy uses high energy x-rays to damage tumor cells.

PURPOSE: Randomized phase III trial to compare the effectiveness of conventional radiation therapy with high-dose radiation therapy in treating men with stage I or stage II prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether high-dose radiotherapy using conformal photons with a proton boost produces a 20% increase in the proportion of Stage I/II prostate cancer free from local failure and biochemical relapse at 5 years when compared to results of conventional-dose radiotherapy. II. Determine whether high-dose radiotherapy produces a 33% reduction in the cumulative incidence of a rising PSA (second hormone failure) following hormone therapy given at the time of first PSA/clinical failure when compared with conventional-dose radiotherapy. IV. Assess the relative rectal, bladder, and sexual morbidity of conformal photon doses of 70.2 and 79.2 Gy in these patients. V. Collect, in a prospective manner, paraffin biopsy blocks for subsequent analysis of emerging molecular pathologic predictors of outcome in three patients.

OUTLINE: Randomized study. Arm I: Radiotherapy. Boost to the prostate using high-LET protons followed by irradiation of the prostate, periprostatic tissues, and seminal vesicles using conformal photons with energies greater than 6 MV. Conventional dose. Arm II: Radiotherapy. As in Arm I. High dose.

PROJECTED ACCRUAL: There will be 390 patients accrued into this study over 3 years. An additional 3.5 years will be required for follow-up.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed adenocarcinoma of the prostate Primary tumor confined to prostate TNM clinical Stages T1b-c or T2a-b No T1a No T1b-c tumor with Gleason grade 1-2/5 No Gleason grade 1-2/5 and PSA less than 4 ng/mL Nodes negative on imaging (Nx) or by surgical sampling (N0) PSA no greater than 15 ng/mL Treatment must begin within 28 days after randomization

PATIENT CHARACTERISTICS: Age: Any age Performance status: Karnofsky 70%-100% Life expectancy: Greater than 10 years Other: No major medical or psychiatric illness that precludes protocol entry No prior or concurrent second malignancy within 5 years except basal cell skin cancer

PRIOR CONCURRENT THERAPY: No prior treatment for prostate cancer

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 1996-01; Study Completion 2005-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony L. Zietman, MD, Study Chair — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Loma Linda University Medical Center, Loma Linda, California
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts

REFERENCES:
- [Result] Coen JJ, Zietman AL, Rossi CJ, Grocela JA, Efstathiou JA, Yan Y, Shipley WU. Comparison of high-dose proton radiotherapy and brachytherapy in localized prostate cancer: a case-matched analysis. Int J Radiat Oncol Biol Phys. 2012 Jan 1;82(1):e25-31. doi: 10.1016/j.ijrobp.2011.01.039. Epub 2011 Apr 4. PMID 21470787
- [Result] Nguyen PL, Chen RC, Hoffman KE, Trofimov A, Efstathiou JA, Coen JJ, Shipley WU, Zietman AL, Talcott JA. Rectal dose-volume histogram parameters are associated with long-term patient-reported gastrointestinal quality of life after conventional and high-dose radiation for prostate cancer: a subgroup analysis of a randomized trial. Int J Radiat Oncol Biol Phys. 2010 Nov 15;78(4):1081-5. doi: 10.1016/j.ijrobp.2009.09.015. Epub 2010 Mar 6. PMID 20207497
- [Result] Zietman AL, Bae K, Slater JD, Shipley WU, Efstathiou JA, Coen JJ, Bush DA, Lunt M, Spiegel DY, Skowronski R, Jabola BR, Rossi CJ. Randomized trial comparing conventional-dose with high-dose conformal radiation therapy in early-stage adenocarcinoma of the prostate: long-term results from proton radiation oncology group/american college of radiology 95-09. J Clin Oncol. 2010 Mar 1;28(7):1106-11. doi: 10.1200/JCO.2009.25.8475. Epub 2010 Feb 1. PMID 20124169
- [Result] Rossi CJ, Zietman AL, DeSilvio M, et al.: A randomized trial comparing conventional dose (70.2GyE) and high-dose (79.2GyE) conformal radiation in early stage adenocarcinoma of the prostate: results of an interim analysis of PROG 95-09. [Abstract] American Society of Clinical Oncology 2005 Prostate Cancer Symposium, 17-19 February 2005, Orlando, Florida. A-58, 2005.
- [Result] Zietman AL, DeSilvio ML, Slater JD, Rossi CJ Jr, Miller DW, Adams JA, Shipley WU. Comparison of conventional-dose vs high-dose conformal radiation therapy in clinically localized adenocarcinoma of the prostate: a randomized controlled trial. JAMA. 2005 Sep 14;294(10):1233-9. doi: 10.1001/jama.294.10.1233. PMID 16160131
- [Result] Zietman AL, DeSilvio M, Slater JD, et al.: A randomized trial comparing conventional dose (70.2GyE) and high-dose (79. 2GyE) conformal radiation in early stage adenocarcinoma of the prostate: results of an interim analysis of PROG 95-09. [Abstract] Int J Radiat Oncol Biol Phys 60 (Suppl 1): A-4, S131, 2004.